CLINICAL TRIAL: NCT04199702
Title: Feasibility and Safety of Same Day Discharge afTer Atrial Fibrillation Ablation
Acronym: FAST-AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not enroll any patients due to lack of resources.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Moussa C Mansour, PI, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019P003413
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Same day discharge (Other)
  Interventions: Other: Same day discharge

INTERVENTIONS:
Other: Same day discharge — Patients will be discharged the same day they undergo catheter ablation of atrial fibrillation.

SUMMARY:
Catheter ablation with pulmonary vein (PV) isolation is a commonly performed strategy employed for the treatment of atrial fibrillation. The conventional approach for post-procedure care has been for the patient to stay overnight and be discharged the next day. However, the overall incidence of procedure related complications of catheter ablation for atrial fibrillation in high volume centers is low. New technologies have been introduced and improve the safety of the ablation procedure. Discharging patients the same day after ablation is a practice that's currently followed by many centers in the United States and abroad. The investigators' hypothesis is that the currently available advanced technologies allow for the same-day safe discharge of patients after catheter ablation. The investigators propose a prospective single-arm study to evaluate the feasibility and safety of the same-day discharge after AF ablation at MGH. The protocol of same-day discharge will include the use of a commercially available venous closure device, early ambulation, bed-side echocardiogram, and follow-up phone calls at day 1 and 3 post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 - Age < 75 yr
* Documentation of atrial fibrillation (AF) or atypical atrial flutter
* All patients must understand and adhere to the requirements of the study and be willing to comply with the post study follow-up requirements

Exclusion Criteria:

* Heart failure with reduced ejection fraction less than 40%
* Any reversible cause of AF (post-surgery, thyroid disorder, etc.)
* INR > 4.0 at the time of the procedure
* Mental impairment precluding verbal consent or completing follow up
* Patients with any other significant uncontrolled or unstable medical condition
* Women who are known to be pregnant or have had a positive β-HCG test within 7 days prior to procedure
* Presence of left atrial thrombus
* Patients with prior prostate hypertrophy or bladder surgery
* BMI > 40 or BMI <20
* Patients with h/o symptomatic heart failure
* Patients with severe aortic stenosis (AS) or severe mitral regurgitation (MR)
* Patients who require femoral arterial line for blood pressure monitoring

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The rate of successful same day discharge after AF ablation procedure | Day of the AF ablation procedure
  The rate of successful same day discharge after AF ablation procedure in more than 80% of cases that undergo the AF ablation procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States